CLINICAL TRIAL: NCT00499512
Title: Evaluation of the Role of Spirituality in Coping With and Surviving Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Role of Spirituality in Coping and Surviving With Ovarian Cancer, Primary Peritoneal or Fallopian Tube Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: The Blanton Davis Ovarian Cancer Research Program (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2004-0283
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Spirituality; Religion; Quality of Life; Questionnaire; Survey
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spirituality Questionnaire: Patients with newly diagnosed ovarian, primary peritoneal, or fallopian tube cancer.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires that ask questions about religion, spirituality, and decisions about treatment at three points (at time of diagnosis, end of primary chemotherapy, and one year later).
  Other Names: Survey

SUMMARY:
The goal of this psychosocial research study is to examine and explain the influence of spirituality on patients with ovarian, primary peritoneal or fallopian tube cancer.

DETAILED DESCRIPTION:
Little is known about the role a patient's spirituality plays in their quality of life. This study consists of a series of questionnaires that ask questions about religion, spirituality, and decisions about treatment.

All patients with newly diagnosed ovarian, primary peritoneal or fallopian tube cancer who come to the Department of Gynecologic Oncology at M. D. Anderson and affiliated clinics for care will be offered study participation.

Patients will be asked to complete a series of questionnaires at specific times: at the time of diagnosis (before their second cycle of therapy begins), at the end of primary chemotherapy, and one year later. The questionnaires should take a total of about 65 minutes to complete, and patients can choose not to answer any question they do not want to answer.

Patients who agree to participate but do not have time to fill out the questionnaires during their visits may return the questionnaire by mail in a pre-stamped envelope.

All participants will be asked to provide the following information: their age, religious preference, race, marital status, date of diagnosis, stage of disease, and their current treatment. This information will be on a data sheet and should take about 5 minutes to complete.

Any collected information will be confidential. Each participant will be given a specific identification number so that confidentiality can be maintained.

This study is partially funded by a research grant from the Blanton Davis Ovarian Cancer Research Program, in Department of Gynecologic Oncology at M. D. Anderson.

This is an investigational study. About 115 participants will be enrolled in this multicenter study.

About 60 participants will be enrolled at MD Anderson. Up to 31 will be enrolled at the Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. All newly diag Stage II-IV ovarian, primary peritoneal or fallopian tube ca patients prior to initiating C2 of chemo. (A pt with synchronous primary endometrial ca, or HX of primary endometrial ca, can participate if these conditions are met: endometrial ca stage not greater than I-B; no more than superficial myometrial invasion, w/o vascular or lymphatic invasion; no poorly differentiated subtypes, incl papillary serous, clear cell or other FIGO G3 lesions; no add'l tx other than req for ovarian, prim. peritoneal or fallopian tube ca is recommended.)
2. Patients who receive neoadjuvant chemotherapy (prior to a planned interval cytoreduction for a suspected ovarian, primary peritoneal or fallopian tube cancer) are also eligible as long as there is pathologic confirmation of cancer prior to study enrollment.

Exclusion Criteria:

1. Patients who do not speak or read English or Spanish.
2. Patients with Stage I ovarian, primary peritoneal or fallopian tube cancer or patients with tumors of low malignant potential or borderline tumors.
3. Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, who do not meet the criteria listed above.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed ovarian, primary peritoneal or fallopian tube cancer.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2005-08-10 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Response to Questionnaire (Spiritual assessments) | From diagnosis to completion of primary therapy and to 1 year after completion of primary therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org